CLINICAL TRIAL: NCT05687721
Title: A Phase II Trial With Copanlisib Plus Avelumab as a Maintenance Therapy for Metastatic Bladder Cancer After Platinum-based Chemotherapy
Brief Title: Copanlisib and Avelumab as a Maintenance Therapy for Advanced Bladder Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study drug is not available.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCA-016-21F; CX002545 (Other Grant/Funding Number: eRA)
Record Dates: First submitted 2023-01-06; First posted 2023-01-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Advanced Urothelial Carcinoma
Keywords: Urinary Bladder Neoplasms; Phosphatidylinositol 3-Kinase; immunotherapy; copanlisib; pembrolizumab; Ureteral Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms | interventions — copanlisib; avelumab

STUDY DESIGN:
Intervention Model Description: This is a single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapeutic arm (Experimental): Copanlisib will be administered through intravenous infusion (IV) at 60 mg on Day 1, 8 and 15, and avelumab will be administered 800 mg IV on Day 1 and 15 of each 4-week treatment cycle for up to 26 cycles
  Interventions: Drug: copanlisib; Drug: Avelumab

INTERVENTIONS:
Drug: copanlisib — intravenous infusion (IV) at 60 mg on Day 1, 8 and 15 of each 4-week treatment cycle for up to 26 cycles
Drug: Avelumab — 800 mg intravenous infusion on Day 1 and 15 of each 4-week treatment cycle for up to 26 cycles

SUMMARY:
Patients with metastatic bladder cancer are usually treated with chemotherapy. If their cancers do not progress after chemotherapy, they can be enrolled into this study and receive a standard-of-care immunotherapy medication named avelumab plus a study drug named copanlisib.

DETAILED DESCRIPTION:
Patients with advanced urothelial cancer will be treated with platinum-based chemotherapy. After chemotherapy, an imaging study will be performed to determine cancer response. If there is no disease progression, patients will be eligible for this study. After informed consent is obtained, patients are enrolled. The treatment include immunotherapy avelumab as the standard of care plus a study medication copanlisib. Both medications are administrated through intravenous infusion. Avelumab wil be given once every two weeks while copanlisib will be administrated on Day 1, 8 and 15 of every 4-week cycle. Patient will be followed up for disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age > 18 years
3. Diagnosis:

   1. Histologically or cytologically confirmed metastatic or recurrent urothelial carcinoma. OR
   2. Documented stage IV disease (T4b, Any N, M0; any T, Any N, M1a-b), or Stage IIIB (T1-T4a, N2-N3, M0), or subset of stage IIIA (T1-T4a, N1, M0)
4. Completed prior first-line platinum-based chemotherapy at least 4 weeks and not more than 10 weeks after the last dose of first line chemotherapy.
5. Patients without progressive disease as per RECIST v1.1 guideline (i.e., with an ongoing CR, PR, or SD) following completion of the first-line chemotherapy.
6. Patient must be appropriate to receive Avelumab maintenance therapy
7. Measurable disease after chemotherapy is not required:

   1. Patients must have had X-rays, CT/ MRI scans, PET or physical examinations completed within 28 days prior to initial administration of study medications.
   2. Patients may have no evidence of disease after platinum-based chemotherapy. These patients will be included in the study for all other analyses except ORR and irORR.
   3. Soft tissue disease that has been radiated within two months prior to registration is not assessable as measurable disease. Soft tissue disease that has been radiated two or more months prior to registration is assessable as measurable disease provided that the lesion has progressed following radiation. As the biology of previously irradiated tumors may be different from non-irradiated tumors, patients must have at least one measurable lesion outside the previously irradiated region in order to be considered to have measurable disease.
8. Tumor samples:

   a.Provision of a recent formalin-fixed, paraffin-embedded (FFPE) tumor tissue block from the most recent primary or metastatic tumor biopsy or resection obtained prior to treatment with first line chemotherapy but within one year of enrollment, with no intervening systemic anti-cancer therapy. If an FFPE tissue block cannot be provided, 15 unstained slides (10 minimum) will be acceptable. If a suitable tissue sample is not otherwise available, then a tissue from a de novo biopsy (core needle or excisional) should have been obtained prior to initiation of this study. However, this biopsy is not required for participation in this trial if he/she meets all other inclusion and exclusion criteria. When patients undergo biopsy, in addition to FFPE preparation, fresh tissue should be sent to VABHS for single-cell RNAseq and T cell receptor sequencing as specified in the addendum.
9. Estimated life expectancy of at least 3 months.
10. Eastern Cooperative Oncology Group (ECOG) performance status (PS) status 2 OR Karnofsky Performance Status scale 60%. For the safety lead-in phase, only patients with PS 0-1 will be included.
11. Adequate bone marrow function, including:

    1. Leukocytes > 3000/mm3
    2. Absolute neutrophil count (ANC) > 1,500/mm3
    3. Platelets > 100,000/mm3
    4. Hemoglobin > 9 g/dL (may have been transfused).
12. Adequate renal function, defined as estimated creatinine clearance 20 mL/minute as calculated using the Cockcroft-Gault equation. It has been shown that creatinine clearance 15 ml/minute did not significantly affect the pharmacokinetics of copanlisib.
13. Adequate liver function, including:

    b.Total serum bilirubin 1.5 x upper limit of normal (ULN) c.Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 2.5 x ULN d.Total serum bilirubin < 3 x ULN for patients with Gilbert's syndrome or for patients with cholestasis due to compressive adenopathy of the hepatic hilum
14. Serum pregnancy test (for females of childbearing potential) negative at screening.
15. Male patients able to father children and female patients of childbearing potential and at risk for pregnancy must agree to use 2 highly effective methods of contraception throughout the study and for at least 60 days after the last dose of assigned treatment.
16. Evidence of a signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
17. Patients who are willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
18. Controlled diabetes A1c < 8.5%. For patients with newly diagnosed diabetes mellitus that cannot meet protocol requirements, a single rescreening (which includes all screening procedures) should be performed when the patient's diabetes is controlled and can meet protocol requirement for HbA1c).
19. Controlled arterial hypertension (per investigator assessment

Exclusion Criteria:

1. Patients whose disease progressed by RECIST v1.1 on or after first-line platinum-based chemotherapy for urothelial cancer.
2. Patients who have had a major surgery within 4 weeks or major radiation therapy within 2 weeks prior to randomization. Prior palliative radiotherapy is permitted, provided it has been completed at least 48 hours prior to entering the study.
3. Patients who are receiving any other investigational agent within the preceding 4 weeks. Observational studies are permitted.
4. Prior treatment with a Phosphoinositide 3-kinase inhibitor.
5. Prior therapy with anti-PD1/PD-L1 monoclonal antibody for aBC. However, prior treatment with adjuvant nivolumab is allowed if it was discontinued over 12 months prior to the start of this trial.
6. Patients with known symptomatic central nervous system (CNS) metastases requiring steroids. These patients have poor prognosis and often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events. Patients with previously diagnosed CNS metastases are eligible if the participants have completed the treatment and have recovered from the acute effects of radiation therapy or surgery prior to treatment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks, and are neurologically stable.
7. Diagnosis of any other malignancy in past 3 years, except for adequately treated basal cell or squamous cell skin cancer, other Stage 0 or Stage 1 cancers, or incidental finding of prostate cancer during cystoprostatectomy.
8. Patients with symptomatic metastatic cancer, such as moderate to severe pain, impaired organ function or spinal cord compression.
9. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
10. Known severe hypersensitivity reactions to monoclonal antibodies (Grade > 3), any history of anaphylaxis, or uncontrolled asthma (i.e., 3 or more features of asthma system controlled per the Global Initiative for Asthma 2015)
11. History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
12. HbA1c > 8.5% at Screening
13. Known prior or suspected hypersensitivity to study drugs or any component in the formulations.
14. Current or prior use of immunosuppressive medication within 7 days prior, except the following:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
    2. Systemic corticosteroids at physiologic doses 10 mg/day of prednisone or equivalent
    3. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
15. Patient with a history or concurrent condition of Interstitial Lung Disease.
16. Patients with an active bleeding diathesis.
17. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident (<6 months prior to enrollment), myocardial infraction (<6 months prior to enrollment), unstable angina, congestive heart failure (> New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
18. Active infection requiring systemic therapy.
19. Positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) due to potential pharmacokinetic interactions with copanlisib.
20. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
21. Other severe acute or chronic medical conditions including, but not limited to pneumonitis; psychiatric condition including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
22. Vaccination within 4 weeks of the first dose of study treatment and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated influenza vaccine and COVID-19 vaccines).
23. Pregnant female patients, breastfeeding female patients, female patients of childbearing potential and male patients who are unwilling or unable to use 2 highly effective methods of contraception as outlined in the protocol for the duration of the study and for at least 60 days after the last dose of investigational product
24. History of noncompliance to medical regimens.
25. Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 months into the trial
  The primary endpoint is PFS. PFS is defined as the time between initiation of the avelumab/copanlisib combination and tumor progression or death from any cause, with censoring of patients who are lost to follow-up.

SECONDARY OUTCOMES:
Overall Survival | 24 months
  Overall survival is defined as the length of time from the start of this trial treatment to the time of death from any cause
Objective response rate | 2 months
  Objective response rate is defined as the percentage of patients who have a partial or complete response at any time during this treatment of this trial
Disease-control rate | 2-8 months
  Disease-control rate is defined as the percentage of patients who have a partial or complete response or stable disease at any time during this treatment of this trial
Adverse events | up to 2 years into the study
  Adverse events are defined as any untoward medical occurrence of subjects which does not necessarily have a causal relationship with the treatment

OTHER OUTCOMES:
Molecular Correlative Studies | up to 2 years into the study
  Immune cell infiltration, immune cell activation/exhaustion status, cytokine production and signaling transduction pathways will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Xian Pan, MD PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT05687721/ICF_000.pdf